CLINICAL TRIAL: NCT07015736
Title: Effect of Saccharomyces Boulardii CNCM I-745 on Antibiotic-perturbed Microbiota in Children: RESTORE STUDY
Brief Title: Effects of Saccharomyces Boulardii CNCM I-745 on Antibiotic-Associated Perturbation in Children Treated for Acute Respiratory Infections (RESTORE Study)
Acronym: RESTORE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Professor in Pediatrics, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Restore-V004-2025-6
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Antibiotic Associated Diarrhea; Acute Otitis Media; ACUTE SINUSITIS
Keywords: antibiotic associated diarrhea; probiotic; microbiota; microbiome; Saccharomyces boulardii
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin-Potassium Clavulanate Combination; Suspensions

STUDY DESIGN:
Masking Description: Microbiota analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotic 10 Days Group (Experimental): Amoxicillin-clavulanic acid + S. boulardii for 10 days
  Interventions: Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension; Dietary Supplement: Saccharomyces boulardii CNCM I-745
- Probiotic 21 Days Group (Experimental): Amoxicillin-clavulanic acid for 10 days + S. boulardii for 21 days (overlapping first 10 days)
  Interventions: Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension; Dietary Supplement: Saccharomyces boulardii CNCM I-745
- Antibiotic-Only Group (Experimental): Amoxicillin-clavulanic acid for 10 days (no probiotic)
  Interventions: Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension
- Healthy Control Group (No Intervention): No infection, antibiotics, or probiotics

INTERVENTIONS:
Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension — Standard treatment (50-90 mg/kg/day for 10 days)
  Arms: Antibiotic-Only Group; Probiotic 10 Days Group; Probiotic 21 Days Group
Dietary Supplement: Saccharomyces boulardii CNCM I-745 — Probiotic sachet, twice daily for 10 or 21 days depending on group assignment
  Arms: Probiotic 10 Days Group; Probiotic 21 Days Group

SUMMARY:
This study aims to evaluate the effect of co-administering the probiotic Saccharomyces boulardii CNCM I-745 with amoxicillin-clavulanic acid on the intestinal and nasopharyngeal microbiota in children diagnosed with acute otitis media or acute bacterial sinusitis. The trial will also assess the potential of the probiotic to reduce antibiotic-associated diarrhea (AAD), antibiotic associated microbiota perturbation, and the spread of antibiotic resistance genes (ARGs).

ELIGIBILITY:
Inclusion Criteria

Diagnosed with acute otitis medica or acute rhinosinusitis

No chronic diseases or recent antibiotic/probiotic use (past 8 weeks)

Parental consent obtained

Exclusion Criteria:

Age <4 or >12 years

Chronic illness or GI disorders

History of antibiotic allergy or immunocompromise

Malnutrition or obesity

Recent gastrointestinal surgery

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in intestinal microbiota bacteria composition | 0, 10, 21 and 56 days
  Change in intestinal microbiota bacteria composition with WGS
Potential changes in antibiotic resistant genes (ARGs) | 0, 10, 21, and 56 days of study
  Potential changes in antibiotic resistant genes (ARGs)

SECONDARY OUTCOMES:
Change in intestinal microbiota virome composition | 0, 10, 14, 56 days of study
  Change in intestinal microbiota virome composition
Change in intestinal microbiota mycobiome composition | 0, 10, 14, 21 days of study
  Change in intestinal microbiota mycobiome composition
Changes in nasopharyngeal microbiota composition | 0, 10, 21, 56 days of intervention
  Changes in nasopharyngeal microbiota bacteriaal composition

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Eskisehir Osmangazi University, Eskişehir
  - Acibadem Univsersity Faculty of Medicine, Istanbul
  - Sancaktepe Şehit Prof.Dr. İlhan Varank Training and Research Hospital, Istanbul
  - Şişli Hamidiye Etfal Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No